CLINICAL TRIAL: NCT03638128
Title: Multicenter, Single-arm Open-label Extension Study to Assess Long-term Safety and Efficacy of Current or Prior Treatment With Denosumab in Children/Young Adults With Osteogenesis Imperfecta
Brief Title: Open-label Extension of Study 20130173 of Denosumab in Children and Young Adults With Osteogenesis Imperfecta
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped earlier than planned due to safety concerns about high levels of calcium in the blood of the participants
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170534; 2018-000550-21 (EudraCT Number)
Record Dates: First submitted 2018-06-21; First posted 2018-08-20 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Osteogenesis Imperfecta (OI)
Keywords: OI; Bone.
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Alternative Medications / Observational (Other): Participants who received non-denosumab alternative therapy during the study or who were not receiving any medication at baseline.
  Alternative osteoporosis medication(s) were determined at the investigator's discretion and per standard of care and local guidelines.
  Interventions: Drug: Alternative osteoporosis medications
- Denosumab 1 mg/kg Q6M (Experimental): Participants who received at least 1 dose of 1 mg/kg denosumab administered once every 6 months (Q6M) by subcutaneous injection, but no Q3M denosumab during this study.
  Interventions: Drug: Denosumab
- Denosumab 1 mg/kg Q3M (Experimental): Participants who received at least one dose of 1 mg/kg denosumab administered once every 3 months (Q3M) by subcutaneous injection during this study.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Solution for injection
  Other Names: Prolia
  Arms: Denosumab 1 mg/kg Q3M; Denosumab 1 mg/kg Q6M
Drug: Alternative osteoporosis medications — Alternative osteoporosis medication/s at the discretion of the investigator.
  Arms: Alternative Medications / Observational

SUMMARY:
To evaluate long-term safety of denosumab in children/young adults with pediatric osteogenesis imperfecta (OI) who completed the prior study 20130173 (NCT02352753).

DETAILED DESCRIPTION:
All participants who completed the prior denosumab study 20130173 (NCT02352753) were offered participation in this study (20170534). Participants could continue to receive denosumab once every 3 months (Q3M) or could receive denosumab once every 6 months (Q6M) or off-treatment observation only at the investigator's discretion. The study design allowed subjects to discontinue denosumab, resume denosumab, initiate alternative osteoporosis medication, discontinue alternative osteoporosis medication, or receive no treatment (observation only) at any time. Therefore results of this study were analyzed according to both baseline treatment and subsequent treatment trajectories.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent/assent prior to initiation of any Study 20170534 specific activities/procedures. Subject's legally acceptable representative has provided informed consent when the subject is legally too young to provide informed consent and the subject has provided written assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated.
* Subject is currently/was enrolled in Study 20130173 and

  * completed the 20130173 End of Study (EOS) visit (regardless of completing or ending investigational product early) OR
  * did not reconsent/reassent to transition to 3-month dosing regimen on Study 20130173 OR
  * early terminated from Study 20130173 as a result of meeting bone mineral density (BMD) Z-score investigational product stopping criteria.

Exclusion Criteria:

* Treatment with any prohibited proscribed medications while receiving denosumab. Eligibility into study treatment with alternative osteoporosis medication/s of investigator's choice, follow guidelines per the specific alternative osteoporosis medication/s selected. For subjects off-treatment (observation only), no prohibited medications apply.
* Subjects currently receiving treatment in another investigational device or drug study other than Study 20130173. Other investigational procedures while participating in this study are excluded.
* For subjects expected to receive investigational product (denosumab) at study day 1: Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 5 months after the last dose of denosumab. Females of childbearing potential (Tanner Stage greater than or equal to 2) should only be included in the study after a negative highly sensitive urine or serum pregnancy test. For study treatment with alternative osteoporosis medication/s of investigator's choice, follow guidelines per the specific alternative osteoporosis medication/s selected. For Subjects off-treatment (observation only), no exclusion applies.
* For subjects expected to receive investigational product (denosumab) at study day 1: Female subjects of childbearing potential unwilling to practice true sexual abstinence (refrain from heterosexual intercourse) or use 1 highly effective method of contraception during treatment and for an additional 5 months after the last dose of investigational product (denosumab). For study treatment with alternative osteoporosis medication/s of investigator's choice, follow contraception guidelines per the specific alternative osteoporosis medication/s selected. For subjects not receiving any investigational product (observation only), no contraception required.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (2):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Indiana University - Riley Hospital for Children, Indianapolis, Indiana
- Australia (2):
  - The Childrens Hospital at Westmead, Westmead, New South Wales
  - Perth Childrens Hospital, Nedlands, Western Australia
- Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels, Belgium
- Canada (3):
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Shriners Hospital for Children, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Plzen, Pilsen
  - Thomayerova nemocnice, Prague
- France (2):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Pellegrin, Bordeaux
  - Hopital Necker Enfants Malades, Paris
- Uniklinik Köln, Cologne, Germany
- Semmelweis Egyetem, Budapest, Hungary
- Azienda Ospedaliera Policlinico Umberto I, Roma, Italy
- SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Lodz, Poland
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
- United Kingdom (4):
  - Birmingham Childrens Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Royal Hospital for Children, Glasgow
  - Sheffield Childrens Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 22 centers in North America, Europe, and Australia from July 2018 to March 2022.
  The study was an open-label extension of study 20130173 (NCT02352753). Participants who completed the end of study visit or who withdrew consent or assent to transition to every 3 months (Q3M) dosing regimen in Study 20130173 were offered participation in this study.
Pre-assignment Details: Participants who rolled over into Study 20170534 could continue to receive denosumab Q3M or could receive alternative osteoporosis medication, including commercial denosumab every 6 months (Q6M), or off-treatment observation only at the investigator's discretion. At any time during the study, participants could discontinue, resume, or initiate 1 of the above treatments based on the medical judgment of the investigator and per local standard of care.
Groups:
- Denosumab 1 mg/kg Q6M: Participants who received at least 1 dose of 1 mg/kg denosumab administered once every 6 months (Q6M) administered by subcutaneous injection, but no Q3M denosumab during this study.
Period: Overall Study
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
Started | 21 | 27 | 27
Completed | 5 | 8 | 1
Not Completed | 16 | 19 | 26
Not completed — Withdrawal by Subject | 1 | 7 | 6
Not completed — Sponsor Decision | 15 | 12 | 19
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M | Total
Number analyzed (Participants) | 21 | 27 | 27 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (3.5) | 13.2 (2.5) | 14.3 (4.8) | 13.4 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 13 | 30
  Male | 13 | 18 | 14 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 20 | 27 | 24 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 0 | 2
  White | 20 | 25 | 23 | 68
  Other | 0 | 1 | 1 | 2
  Multiple | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest
Description: A Serious Adverse Event is defined as any untoward medical occurrence that met at least 1 of the following serious criteria:
  * Resulted in death (fatal)
  * Immediately life-threatening
  * Required in-patient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Was a congenital anomaly/birth defect
  * Other medically important serious event that may have jeopardized the participant or require medical or surgical intervention to prevent 1 of the outcomes listed above.
  Adverse events of special interest included hypocalcemia, hypersensitivity, bacterial cellulitis, osteonecrosis of the jaw (ONJ), hypercalcemia, and typical osteogenesis imperfecta (OI) femur fractures.
Time Frame: From enrollment to end of study, including 24 weeks after last dose of denosumab for participants who received denosumab; the maximum time on study was 24 months.
Population: The safety analysis set includes all enrolled participants who provided informed consent/assent, had a non-missing enrollment date, and received at least 1 dose of denosumab during Study 20130173.
Measure: Count of Participants; unit: Participants
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
Number analyzed (Participants) | 21 | 27 | 27
Participants
  Any adverse event | 18 | 22 | 19
  Serious adverse events | 6 | 5 | 6
  Adverse events of special interest | 5 | 5 | 9
  Hypocalcemia | 0 | 0 | 1
  Hypercalcemia | 3 | 4 | 9
  Hypersensitivity | 0 | 0 | 0
  Bacterial cellulitis (skin infection) | 0 | 0 | 0
  Typical osteogenesis imperfecta femur fractures | 2 | 1 | 2
  Positively adjudicated osteonecrosis of the jaw | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Anti-denosumab Antibodies
Description: Blood samples were collected (from denosumab treated participants only) for the measurement of anti-denosumab binding antibodies. Samples positive for anti-denosumab binding antibodies were further tested for neutralizing antibodies.
Time Frame: as for outcome 1
Population: Safety analysis set participants who received at least one dose of denosumab in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
Number analyzed (Participants) | 27 | 27
Participants
  Anti-denosumab binding antibodies | 0 | 0
  Anti-denosumab neutralizing antibodies | 0 | 0

3. Primary Outcome: Number of Participants With Clinical Laboratory Toxicities Grade ≥ 3
Description: Laboratory abnormalities were graded according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0. The grades refer to the severity of the finding:
  Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant; Grade 4 = Life-threatening consequences, urgent intervention indicated.
Time Frame: as for outcome 1
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
Number analyzed (Participants) | 21 | 27 | 27
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Vital Sign Findings
Description: Vital sign measurements included systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature. The investigator assessed vital sign results and determined whether any abnormal changes represented a clinically significant change from the participant's baseline values.
Time Frame: as for outcome 1
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
Number analyzed (Participants) | 21 | 27 | 27
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Metaphyseal Index Z-score Above Age-appropriate Normal Range
Description: Anteroposterior radiographs of both knees (unless prohibited by the presence of hardware such as implants) were used to calculate the metaphyseal index Z-score of each knee in participants with open growth plates; the knee selected for assessment during the study was the knee with the higher Z-score at baseline. The metaphyseal index (MI) was calculated by the central imaging vendor as the ratio of femoral width over distal femoral growth plate width, and the Z-score for each participant, relative to the participant's age as:
  MI Z-score = (participant value - mean)/SD, where mean and standard deviation (SD) are the corresponding values based on a reference population for the participant's age group at the time of the assessment.
  Metaphyseal index Z-score above age-appropriate normal range is defined as a MI Z-score > 2.
Time Frame: Baseline, month 12 and month 24
Population: The metaphyseal analysis set includes participants with open growth plates and no hardware preventing accurate calculation of MI at baseline, and X-ray of the knee at baseline and postbaseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
Number analyzed (Participants) | 3 | 4 | 4
Participants
  Baseline | 2 | 1 | 0
  Month 12 | 2 | 1 | 0
  Month 24: number analyzed (Participants) | 1 | 1 | 0
  Month 24 | 1 | 0 |

6. Primary Outcome: Number of Participants With Abnormal Molar Eruption of the First or Second Molar Based on Radiological Findings
Description: Participants underwent a visual inspection under natural light for the presence of the first and second molars. Participants were referred to a dentist to perform radiographic assessment of the unerupted molar(s) if:
  * A participant was age 7 to 12 years and appeared to have an unerupted upper or lower first molar (ie, not all 4 first molars were visible/detectable).
  * A participant was age 13 years or older and appeared to have an unerupted upper or lower (first or) second molar (ie, not all 4 first molars and all 4 second molars were visible/detectable).
  Abnormal molar eruptions includes the number of participants 7 to 12 years of age with 1st unerupted or partially erupted molars and participants 13 years of age or older with 2nd unerupted or partially erupted molars.
Time Frame: Baseline, month 12, and month 24
Population: Safety analysis set participants with radiologic assessments at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
Number analyzed (Participants) | 19 | 22 | 17
Participants
  Baseline | 2 | 3 | 1
  Month 12: number analyzed (Participants) | 10 | 8 | 6
  Month 12 | 0 | 0 | 2
  Month 24: number analyzed (Participants) | 2 | 8 | 1
  Month 24 | 1 | 1 | 0

7. Primary Outcome: Percent Change From Baseline in Mandibular Shaping Parameters
Description: Lateral cephalogram was performed to enable assessment of mandibular shaping. The lateral cephalogram is a profile X-ray of the skull and soft tissues and is used to assess the relation of the teeth in the jaws, the relation of the jaws to the skull, and the relation of the soft tissues to the teeth and jaws.
  The following anatomical angles and dimensions were measured to evaluate the correct proportions of the mandible and its position relative to the skull/maxilla: Gonial angle; Sella-Nasion-A Point Angle (SNA angle); Sella-Nasion-B Point Angle (SNB angle); and A Point - Nasion-B Point Angle (ANB Angle).
Time Frame: Baseline and month 12 and month 24
Population: Safety analysis set participants with radiologic assessments at baseline and each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
Number analyzed (Participants) | 10 | 15 | 1
percent change
  Gonial angle: month 12: number analyzed (Participants) | 8 | 8 | 1
  Gonial angle: month 12 | 0.5 (2.4) | -1.4 (1.7) | -1.0
  Gonial angle: month 24: number analyzed (Participants) | 2 | 7 | 0
  Gonial angle: month 24 | -2.1 (3.1) | -1.4 (2.2) |
  SNA angle: month 12: number analyzed (Participants) | 8 | 8 | 1
  SNA angle: month 12 | 1.38 (2.09) | 0.37 (2.41) | 0.20
  SNA angle: month 24: number analyzed (Participants) | 2 | 7 | 0
  SNA angle: month 24 | -0.07 (0.73) | -1.70 (1.79) |
  SNB angle: month 12: number analyzed (Participants) | 6 | 8 | 1
  SNB angle: month 12 | 0.98 (1.56) | 1.75 (2.36) | 0.70
  SNB angle: month 24: number analyzed (Participants) | 1 | 4 | 0
  SNB angle: month 24 | 1.28 | -1.60 (3.18) |
  ANB angle: month 12: number analyzed (Participants) | 6 | 8 | 1
  ANB angle: month 12 | -81.06 (199.39) | 127.48 (312.99) | -16.26
  ANB angle: month 24: number analyzed (Participants) | 1 | 4 | 0
  ANB angle: month 24 | -79.69 | 15.65 (84.75) |

8. Secondary Outcome: Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) Z-score
Description: Bone densitometry assessments of the lumbar spine were performed using dual X-ray absorptiometry (DXA).
  The Z-score indicates the number of standard deviations away from the mean of an average person of the same age, sex, race, and weight. A Z-score of 0 is equal to the mean of the matched population, negative Z-scores indicate a BMD lower than the mean of the matched population, and positive Z-scores indicate a higher BMD than that of the matched population. A positive change from baseline indicates an improvement in lumbar spine BMD.
Time Frame: Baseline and months 6, 12, and 24
Population: The DXA analysis set includes all participants with baseline and ≥ 1 postbaseline valid DXA assessments for lumbar spine as provided by the central imaging vendor.
  BMD endpoints were pre-specified to be analyzed for combined treatment groups.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Any Treatment: Participants who were enrolled in the study and received denosumab Q3M or Q6M, alternative treatment or did not receive any treatment.
Arm/Group | Any Treatment
Number analyzed (Participants) | 58
Z-score
  Month 6: number analyzed (Participants) | 29
  Month 6 | -0.11 (0.60)
  Month 12: number analyzed (Participants) | 39
  Month 12 | -0.01 (0.48)
  Month 24: number analyzed (Participants) | 18
  Month 24 | 0.21 (0.49)

9. Secondary Outcome: Change From Baseline in Total Hip BMD Z-score
Description: Bone densitometry assessments of the hip were performed using dual X-ray absorptiometry (DXA).
  The Z-score indicates the number of standard deviations away from the mean of an average person of the same age, sex, race, and weight. A Z-score of 0 is equal to the mean of the matched population, negative Z-scores indicate a BMD lower than the mean of the matched population, and positive Z-scores indicate a higher BMD than that of the matched population. A positive change from baseline indicates an improvement in total hip BMD.
Time Frame: Baseline, months 6, 12, and 24
Population: The DXA analysis set includes all participants with baseline and ≥ 1 postbaseline valid DXA assessments for the total hip as provided by the central imaging vendor.
  BMD endpoints were pre-specified to be analyzed for combined treatment groups.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Any Treatment
Number analyzed (Participants) | 35
Z-score
  Month 6: number analyzed (Participants) | 16
  Month 6 | -0.07 (0.40)
  Month 12: number analyzed (Participants) | 25
  Month 12 | 0.24 (0.42)
  Month 24: number analyzed (Participants) | 15
  Month 24 | 0.50 (0.54)

10. Secondary Outcome: Change From Baseline in Femoral Neck BMD Z-score
Description: Bone densitometry assessments of the femoral neck were performed using dual X-ray absorptiometry (DXA).
  The Z-score indicates the number of standard deviations away from the mean of an average person of the same age, sex, race, and weight. A Z-score of 0 is equal to the mean of the matched population, negative Z-scores indicate a BMD lower than the mean of the matched population, and positive Z-scores indicate a higher BMD than that of the matched population. A positive change from baseline indicates an improvement in femoral neck BMD.
Time Frame: Baseline and months 6, 12, and 24
Population: The DXA analysis set includes all participants with baseline and ≥ 1 postbaseline valid DXA assessments for the femoral neck as provided by the central imaging vendor.
  BMD endpoints were pre-specified to be analyzed for combined treatment groups.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Any Treatment
Number analyzed (Participants) | 35
Z-score
  Month 6: number analyzed (Participants) | 16
  Month 6 | 0.08 (0.44)
  Month 12: number analyzed (Participants) | 25
  Month 12 | 0.24 (0.39)
  Month 24: number analyzed (Participants) | 15
  Month 24 | 0.45 (0.58)

ADVERSE EVENTS:
Time Frame: From enrollment to end of study, including 24 weeks after last dose of denosumab for participants who received denosumab; the maximum time on study was 24 months.
Arm/Group | Alternative Medications / Observational | Denosumab 1 mg/kg Q6M | Denosumab 1 mg/kg Q3M
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 6/21 | 5/27 | 6/27
Other Adverse Events (participants affected / at risk) | 15/21 | 21/27 | 13/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alternative Medications / Observational (N=21) | Denosumab 1 mg/kg Q6M (N=27) | Denosumab 1 mg/kg Q3M (N=27)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Surgical failure (General disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 5
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alternative Medications / Observational (N=21) | Denosumab 1 mg/kg Q6M (N=27) | Denosumab 1 mg/kg Q3M (N=27)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2
COVID-19 (Infections and infestations) | 1 | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 7 | 0
Headache (Nervous system disorders) | 3 | 1 | 2
Hypercalciuria (Renal and urinary disorders) | 11 | 15 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT03638128/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03638128/SAP_001.pdf